CLINICAL TRIAL: NCT01907113
Title: Pharmacokinetics, Pharmacodynamics, Safety and Tolerability of a Single 50 mg Dose of BI 10773 in Patients With Different Degrees of Renal Impairment in Comparison to Subjects With Type 2 Diabetes and Normal Renal Function in a Monocentric, Open-label, Parallel-group, Phase 1 Trial
Brief Title: Pharmacokinetics, Pharmacodynamics, Safety and Tolerability of BI 10773 in Type II Diabetes Patients With Different Degrees of Renal Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1245.12; 2008-006086-86 (EudraCT Number: EudraCT)
Record Dates: First submitted 2013-07-15; First posted 2013-07-24 (Estimated); Results first posted 2014-07-14 (Estimated); Last update posted 2014-07-14 (Estimated); Status verified 2014-07

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — empagliflozin

ARMS (5):
- BI 10773 / Group 2 (Experimental): Single Dose Administration (type 2 diabetes and mild renal impairment)
  Interventions: Drug: BI 10773
- BI 10773 / Group 3 (Experimental): Single Dose Administration (type 2 diabetes and moderate renal impairment)
  Interventions: Drug: BI 10773
- BI 10773 / Group 4 (Experimental): Single Dose Administration (severe renal impairment 8)
  Interventions: Drug: BI 10773
- BI 10773 / Group 5 (Experimental): Single Dose Administration (kidney failure)
  Interventions: Drug: BI 10773
- BI 10773 / Group 1 (Experimental): Single Dose Administration (type 2 diabetes and normal renal function)
  Interventions: Drug: BI 10773

INTERVENTIONS:
Drug: BI 10773 — oral administration
  Arms: BI 10773 / Group 2
Drug: BI 10773 — oral administration
  Arms: BI 10773 / Group 1
Drug: BI 10773 — oral administration
  Arms: BI 10773 / Group 3
Drug: BI 10773 — oral administration
  Arms: BI 10773 / Group 4
Drug: BI 10773 — oral administration
  Arms: BI 10773 / Group 5

SUMMARY:
Assessment of the effect of normal and impaired kidney function on the pharmacokinetics, pharmacodynamics and safety of BI 10773

ELIGIBILITY:
Inclusion criteria:

1. Male and female subjects with type 2 diabetes
2. Renally impaired male or female subjects
3. Age 18 - 75 years
4. BMI 18 - 34 kg/m2, at least 45 kg for females (Body Mass Index)
5. Signed and dated written informed consent

Exclusion criteria:

1. Significant gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders as judged by the investigator.
2. Relevant gastrointestinal tract surgery
3. Diseases of the central nervous system (such as epilepsy, seizures) or psychiatric disorders or relevant neurological disorders
4. History of relevant orthostatic hypotension, fainting spells or blackouts; systolic blood pressure < 100 or > 160 mm Hg, diastolic blood pressure < 60 or > 100 mm Hg, pulse rate < 50 or > 100 1/min
5. Chronic or relevant acute infections
6. History of allergy/hypersensitivity (including drug allergies) that are deemed relevant to the trial as judged by the investigator
7. Use within 10 days prior to administration or during the trial of drugs which might reasonably influence the results of the trial based on the knowledge at the time of protocol preparation. Co medication known to inhibit or induce P-glycoprotein or CYP3A is not allowed. Inhibitors of P-glycoprotein or CYP3A (cytochrom P3A) are e.g.

   * protease inhibitors, (e.g. ritonavir, lopinavir nelfinavir)
   * azole antimycotics, (itraconazole, ketoconazole, miconazole)
   * macrolid antibiotics, (clarithromycin, erythromycin)
   * amiodarone, cimetidine, diltiazem, fluvoxamine, mibefradil, nefazodone, verapamil, tacrolimus, quinidine, reserpine, cyclosporine A Inducers of P-gp or CYP3A are e.g. carbamazepine, phenobarbital, phenytoin, rifabutin, ri-fampin, St. John's wort, troglitazone. In dubious cases, a case by case decision will be made after consultation with the sponsor.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-07; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (2):
- Germany (2):
  - 1245.12.1 Boehringer Ingelheim Investigational Site, Kiel
  - 1245.12.2 Boehringer Ingelheim Investigational Site, Neuss

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted in two trial centres as an open-label, parallel group design with one treatment period.
  The trial was performed in 40 male and female patients who were assigned to five treatment groups according to their creatinine clearance.
Groups:
- Normal Renal Function: Patients with type 2 diabetes and normal renal function. Normal renal function was defined as a Glomerular filtration rate of more than 90 mL/min/1.73 m².
  Patients were administered once with 50 mg of Empagliflozin as a single dose by oral administration.
- Mild Renal Impairment: Patients with type 2 diabetes and mild renal impairment. Mild renal impairment was defined as a Glomerular filtration rate of 60-89 mL/min/1.73 m².
  Patients were administered once with 50 mg of Empagliflozin as a single dose by oral administration.
- Moderate Renal Impairment: Patients with type 2 diabetes and moderate renal impairment. Moderate renal impairment was defined as a Glomerular filtration rate of 30-59 mL/min/1.73 m².
  Patients were administered once with 50 mg of Empagliflozin as a single dose by oral administration.
- Severe Renal Impairment: Patients with severe renal impairment. Severe renal impairment was defined as a Glomerular filtration rate of less than 30 mL/min/1.73 m².
  Patients were administered once with 50 mg of Empagliflozin as a single dose by oral administration.
- Kidney Failure: Patients with kidney failure, i.e. patients requiring dialysis. Patients were administered once with 50 mg of Empagliflozin as a single dose by oral administration.
Period: Overall Study
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment | Kidney Failure
Started | 8 | 9 | 7 | 8 | 8
Completed | 8 | 9 | 7 | 8 | 8
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The treated set included all patients who were dispensed study medication and were documented to have at least one dose of investigational treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment | Kidney Failure | Total
Number analyzed (Participants) | 8 | 9 | 7 | 8 | 8 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.5 (11.7) | 60.0 (8.8) | 63.1 (9.5) | 56.0 (12.9) | 45.8 (12.0) | 55.8 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 3 | 1 | 4 | 21
  Male | 1 | 3 | 4 | 7 | 4 | 19

OUTCOME MEASURES:

1. Primary Outcome: AUC0-∞ (Area Under the Concentration Time Curve of the Analyte in Plasma Over the Time Interval From 0 to Infinity)
Description: Area under the concentration time curve of the analyte in plasma over the time interval from 0 to infinity. The areas under the curve were calculated using the linear up/log down algorithm. If a drug concentration was equal to or higher than the preceding concentration, the linear trapezoidal method was used. If the drug concentration was smaller than the preceding concentration, the logarithmic method was used.
Time Frame: 1 hour (h) before drug administration and 0:20, 0:40, 1:00, 1:30, 2:00, 2:30, 3:00, 4:00, 6:00, 8:00, 10:00, 12:00, 14:00, 24:00, 36:00. 48:00, 72:00, 96:00 h after drug administration
Population: The PK analysis set (PKS) included all evaluable patients in the treated set who provided at least one observation for at least one primary (PK) endpoint without important protocol violations relevant to the evaluation of PK.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment | Kidney Failure
Number analyzed (Participants) | 8 | 9 | 7 | 8 | 8
nmol*h/L | 10500 (17.6) | 12400 (21.6) | 12600 (27.1) | 17500 (18.9) | 15600 (38.6)
Statistical Analysis 1: Comparison: Normal Renal Function vs Mild Renal Impairment; No formal testing, investigation of relative bioavailability; Test type: Non-Inferiority or Equivalence — Ratio calculated as mild renal function divided by normal renal function; ANOVA; Based on ANOVA with fixed effect for treatment (corresponding to renal impairment status); Geometric mean ratio = 118.24, 90% CI 2-sided [96.17 to 145.38], Standard Deviation 25.6 — Standard deviation is actually the geometric Coefficient of Variation [%]
Statistical Analysis 2: Comparison: Normal Renal Function vs Moderate Renal Impairment; No formal testing, investigation of relative bioavailability; Test type: Non-Inferiority or Equivalence — Ratio calculated as moderate renal function divided by normal renal function; ANOVA; Based on ANOVA with fixed effect for treatment (corresponding to renal impairment status); Geometric mean ratio = 119.94, 90% CI 2-sided [96.25 to 149.47], Standard Deviation 25.6 — Standard deviation is actually the geometric Coefficient of Variation [%]
Statistical Analysis 3: Comparison: Normal Renal Function vs Severe Renal Impairment; No formal testing, investigation of relative bioavailability; Test type: Non-Inferiority or Equivalence — Ratio calculated as severe renal function divided by normal renal function; ANOVA; Based on ANOVA with fixed effect for treatment (corresponding to renal impairment status); Geometric mean ratio = 166.29, 90% CI 2-sided [134.44 to 205.68], Standard Deviation 25.6 — Standard deviation is actually the geometric Coefficient of Variation [%]
Statistical Analysis 4: Comparison: Normal Renal Function vs Kidney Failure; No formal testing, investigation of relative bioavailability; Test type: Non-Inferiority or Equivalence — Ratio calculated as kidney failure divided by normal renal function; ANOVA; Based on ANOVA with fixed effect for treatment (corresponding to renal impairment status); Geometric mean ratio = 148.29, 90% CI 2-sided [119.89 to 183.42], Standard Deviation 25.6 — Standard deviation is actually the geometric Coefficient of Variation [%]

2. Primary Outcome: Cmax (Maximum Concentration of the Analyte in Plasma)
Description: Maximum concentration of Empagliflozin in plasma
Time Frame: as for outcome 1
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment | Kidney Failure
Number analyzed (Participants) | 8 | 9 | 7 | 8 | 8
nmol/L | 1210 (24.1) | 1430 (33.1) | 1230 (30.9) | 1450 (33.0) | 1250 (25.9)
Statistical Analysis 1: Comparison: Normal Renal Function vs Mild Renal Impairment; No formal testing, investigation of relative bioavailability; Test type: Non-Inferiority or Equivalence — Ratio calculated as mild renal function divided by normal renal function; ANOVA; Based on ANOVA with fixed effect for treatment (corresponding to renal impairment status); Geometric mean ratio = 118.83, 90% CI 2-sided [93.62 to 150.84], Standard Deviation 29.7 — Standard deviation is actually the geometric Coefficient of Variation [%]
Statistical Analysis 2: Comparison: Normal Renal Function vs Moderate Renal Impairment; No formal testing, investigation of relative bioavailability; Test type: Non-Inferiority or Equivalence — Ratio calculated as moderate renal function divided by normal renal function; ANOVA; Based on ANOVA with fixed effect for treatment (corresponding to renal impairment status); Geometric mean ratio = 102.27, 90% CI 2-sided [79.33 to 131.85], Standard Deviation 29.7 — Standard deviation is actually the geometric Coefficient of Variation [%]
Statistical Analysis 3: Comparison: Normal Renal Function vs Severe Renal Impairment; No formal testing, investigation of relative bioavailability; Test type: Non-Inferiority or Equivalence — Ratio calculated as severe renal function divided by normal renal function; ANOVA; Based on ANOVA with fixed effect for treatment (corresponding to renal impairment status); Geometric mean ratio = 120.68, 90% CI 2-sided [94.42 to 154.25], Standard Deviation 29.7 — Standard deviation is actually the geometric Coefficient of Variation [%]
Statistical Analysis 4: Comparison: Normal Renal Function vs Kidney Failure; No formal testing, investigation of relative bioavailability; Test type: Non-Inferiority or Equivalence — Ratio calculated as kidney failure divided by normal renal function; ANOVA; Based on ANOVA with fixed effect for treatment (corresponding to renal impairment status); Geometric mean ratio = 103.75, 95% CI 2-sided [81.18 to 132.61], Standard Deviation 29.7 — Standard deviation is actually the geometric Coefficient of Variation [%]

3. Secondary Outcome: Time to Maximum Concentration of the Analyte in Plasma
Description: Time from last dosing to maximum concentration of Empagliflozin in plasma (tmax)
Time Frame: 1 h before drug administration and 0:20, 0:40, 1:00, 1:30, 2:00, 2:30, 3:00, 4:00, 6:00, 8:00, 10:00, 12:00, 14:00, 24:00, 36:00. 48:00, 72:00, 96:00 h after drug administration
Population: PKS
Measure: Median (Full Range); unit: h
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment | Kidney Failure
Number analyzed (Participants) | 8 | 9 | 7 | 8 | 8
h | 1.00 [1.00 to 3.00] | 2.50 [2.00 to 4.00] | 2.00 [1.50 to 3.00] | 2.00 [0.67 to 4.00] | 2.50 [1.50 to 3.00]

4. Secondary Outcome: Half-life and Mean Residence Time of the Analyte in Plasma
Description: Terminal half-life of Empagliflozin (t1/2) and Mean residence time of Empagliflozin in the body
Time Frame: as for outcome 3
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment | Kidney Failure
Number analyzed (Participants) | 8 | 9 | 7 | 8 | 8
h
  Terminal half-life | 17.4 (57.4) | 19.3 (81.6) | 19.5 (63.9) | 22.5 (74.3) | 18.5 (62.6)
  Mean residence time | 13.1 (37.4) | 15.7 (44.6) | 18.4 (52.7) | 22.2 (57.6) | 19.8 (51.2)

5. Secondary Outcome: Terminal Rate Constant in Plasma
Description: Terminal rate constant in plasma (Lz)
Time Frame: as for outcome 3
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/h
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment | Kidney Failure
Number analyzed (Participants) | 8 | 9 | 7 | 8 | 8
1/h | 0.0398 (57.4) | 0.0360 (81.6) | 0.0355 (63.9) | 0.0308 (74.3) | 0.0375 (62.6)

6. Secondary Outcome: Apparent Clearance of the Analyte in the Plasma After Extravascular Administration
Description: Apparent clearance of the analyte in the plasma after extravascular administration
Time Frame: as for outcome 3
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/min
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment | Kidney Failure
Number analyzed (Participants) | 8 | 9 | 7 | 8 | 8
mL/min | 176 (17.6) | 149 (21.6) | 147 (27.1) | 106 (18.9) | 119 (38.6)

7. Secondary Outcome: Apparent Volume of Distribution During the Terminal Phase Lz
Description: Apparent volume of distribution during the terminal phase Lz
Time Frame: as for outcome 3
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment | Kidney Failure
Number analyzed (Participants) | 8 | 9 | 7 | 8 | 8
L | 266 (55.1) | 248 (76.3) | 248 (55.5) | 206 (78.0) | 190 (45.1)

8. Secondary Outcome: AUC0-tz (Area Under the Concentration-time Curve of the Analyte in Plasma Over the Time Interval From 0 to the Time of the Last Quantifiable Data Point)
Description: Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the time of the last quantifiable data point. The areas under the curve were calculated using the linear up/log down algorithm. If a drug concentration was equal to or higher than the preceding concentration, the linear trapezoidal method was used. If the drug concentration was smaller than the preceding concentration, the logarithmic method was used.
Time Frame: as for outcome 3
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment | Kidney Failure
Number analyzed (Participants) | 8 | 9 | 7 | 8 | 8
nmol*h/L | 10300 (17.5) | 12100 (20.9) | 12100 (24.4) | 16500 (19.9) | 14900 (34.4)

9. Secondary Outcome: Ae0-96 (Amount of Analyte That is Eliminated in Urine Over the Time Interval 0 to 96 h)
Description: Amount of analyte that is eliminated in urine over the time interval 0-96 hours.
Time Frame: 24-0 h before drug administration and 0-4, 4-8, 8-12, 12-24, 24-36, 36-48, 48-72, 72-96 hours after drug administration
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment | Kidney Failure
Number analyzed (Participants) | 8 | 9 | 7 | 8 | 5
nmol | 17300 (26.1) | 12100 (43.8) | 6840 (85.5) | 3730 (49.3) | 300 (117)

10. Secondary Outcome: fe0-96 (Fraction of Analyte Excreted Unchanged in Urine From Time Points 0 to 96 Hours)
Description: Fraction of analyte excreted unchanged in urine from time point 0-96 hours.
Time Frame: 24-0 h before drug administration and 0-4, 4-8, 8-12, 12-24, 24-36, 36-48, 48-72, 72-96 hours after drug administration
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage of analyte
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment | Kidney Failure
Number analyzed (Participants) | 8 | 9 | 7 | 8 | 5
percentage of analyte | 15.6 (26.1) | 10.9 (43.8) | 6.16 (85.5) | 3.36 (49.3) | 0.271 (117)

11. Secondary Outcome: Renal Clearance of the Analyte in Plasma After Extravascular Administration
Description: Renal Clearance of the Analyte in Plasma After Extravascular Administration for time interval 0-96 hours.
Time Frame: 24-0 h before drug administration and 0-4, 4-8, 8-12, 12-24, 24-36, 36-48, 48-72, 72-96 hours after drug administration
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/min
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment | Kidney Failure
Number analyzed (Participants) | 8 | 9 | 7 | 8 | 5
mL/min | 28.0 (19.5) | 16.7 (53.7) | 9.39 (87.9) | 3.70 (38.5) | 0.349 (188)

12. Secondary Outcome: %AUCtz-∞ (Percentage of Area Under the Concentration-time Curve of the Analyte in Plasma Over the Time Interval From the Time of the Last Quantifiable Data Point Extrapolated to Infinity)
Description: Percentage of area under the concentration-time curve of the analyte in plasma over the time interval from the time of the last quantifiable data point extrapolated to infinity
Time Frame: as for outcome 3
Population: PKS
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percent
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment | Kidney Failure
Number analyzed (Participants) | 8 | 9 | 7 | 8 | 8
percent | 0.869 (225) | 1.07 (243) | 1.21 (223) | 1.78 (334) | 1.14 (330)

13. Secondary Outcome: Plasma Protein Binding
Description: Plasma protein binding is the percent of analyte binding to the plasma protein, pre-dose plasma samples were spiked with Empa 1000 nmol/L.
  The standard deviation is actually the coefficient of variation.
Time Frame: 1 h before drug administration and 1:30 and 3:00 h after drug administration
Population: PKS
Measure: Mean (Standard Deviation); unit: percentage of plasma protein binding
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment | Kidney Failure
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8
percentage of plasma protein binding
  Pre-dose | 83.61 (1.10) | 82.72 (3.36) | 81.29 (2.48) | 79.98 (2.42) | 81.08 (1.54)
  1:30 h after dosing | 85.18 (1.91) | 83.70 (2.49) | 82.68 (2.76) | 81.02 (1.73) | 81.09 (1.94)
  3:00 h after dosing | 83.94 (1.88) | 83.18 (2.58) | 81.90 (1.69) | 80.38 (1.61) | 80.32 (2.00)

14. Secondary Outcome: Total Urinary Glucose Excretion (UGE)
Description: Change from baseline in total urinary glucose excretion
Time Frame: 24-0 h before drug administration and 0-4, 4-8, 8-12, 12-24, 24-36, 36-48, 48-72, 72-96 hours after drug administration (Interval 24-0 h before drug administration only for baseline UGE)
Population: The UGE analysis set included all patients in the treated set who provided the baseline value from 0 to 24 hours before drug administration and the value for urinary glucose excretion from 0 to 24 hours after drug administration without important protocol violations relevant to the evaluation of Pharmacodynamics.
Measure: Mean (Standard Error); unit: mg
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment | Kidney Failure
Number analyzed (Participants) | 8 | 7 | 5 | 6 | 5
mg | 97643 (7204) | 61590 (6892) | 55674 (16891) | 18251 (3925) | 779 (904)

15. Secondary Outcome: Safety: Physical Examination, Vital Signs, ECG and Laboratory Measurements
Description: Number of participants with clinically relevant findings in physical examination, Vital Signs, Clinically Significant Abnormalities in Electrocardiogram (ECG) and Significant Changes from Baseline Laboratory Measurements
Time Frame: Drug administration until end-of-study-examination, 5 days
Population: Treated set
Measure: Number; unit: participants
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment | Kidney Failure
Number analyzed (Participants) | 8 | 9 | 7 | 8 | 8
participants
  Physical examination | 0 | 0 | 0 | 0 | 0
  Vital signs | 0 | 0 | 0 | 0 | 0
  ECG | 0 | 0 | 0 | 0 | 0
  Laboratory Measurements | 0 | 0 | 0 | 0 | 0

16. Secondary Outcome: Assessment of Tolerability by Investigator
Description: Tolerability was assessed by the investigator based on adverse events and the laboratory evaluation.
Time Frame: Drug administration until end-of-study-examination, 5 days
Population: Treated set
Measure: Number; unit: participants
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment | Kidney Failure
Number analyzed (Participants) | 8 | 9 | 7 | 8 | 8
participants
  Good | 8 | 9 | 7 | 8 | 8
  Satisfactory | 0 | 0 | 0 | 0 | 0
  Not satisfactory | 0 | 0 | 0 | 0 | 0
  Bad | 0 | 0 | 0 | 0 | 0
  Not assessable | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From drug administration until end of trial examination, 5 days
Arm/Group | Normal Renal Function | Mild Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment | Kidney Failure
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/9 | 0/7 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 1/8 | 0/9 | 1/7 | 0/8 | 2/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Normal Renal Function (N=8) | Mild Renal Impairment (N=9) | Moderate Renal Impairment (N=7) | Severe Renal Impairment (N=8) | Kidney Failure (N=8)
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Erythema (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.